CLINICAL TRIAL: NCT02652442
Title: Vestibular Rehabilitation and Otolith Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C2058-P
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Dizziness
Keywords: dizziness; postural balance; rehabilitation
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Intervention Model Description: To determine optimal stimulus parameters for off-axis rotation (OAR), participants progressed through the study starting with off-axis distance (3.5 vs 7.0 cm), off-axis duration (1 vs 3 minutes) and finally training schedule (daily vs biweekly). SVV was measured immediately before and after training.
  To determine optimal distance, OAR was first performed at 3.5 cm and then 7.0 cm off-axis for 1 minute and the change in SVV compared. Participants trained daily for 5 consecutive days at 3.5 cm followed by a washout period of two weeks, then trained at 7.0 cm.
  To determine optimal duration, participants were rotated at 3.5 cm off-axis (determined to be optimal) for 3 minutes and the change in SVV was compared to 3.5 cm off-axis for 1 minute.
  To determine optimal training schedule, participants were rotated at 3.5 cm off-axis for 3 minutes (determined to be optimal) on a biweekly schedule for a total of 5 sessions and change in SVV was compared to the daily training schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Centrifugation Parameters (Experimental): Three experiments were performed to identify optimal centrifugation parameters: (1) distance off-axis (3.5 vs 7 cm); (2) duration (1 min vs 3 mins); (3) schedule (daily vs biweekly). The comparisons were all within subjects; i.e., each subject was tested systematically for each centrifugation parameter under both conditions. The change in the outcome measure SVV (from pre- to post-off-axis rotation) for each condition (e.g., 3.5 vs 7 cm) within a parameter was compared.
  Interventions: Behavioral: Centrifugation Distance; Behavioral: Centrifugation Duration; Behavioral: Centrifugation Schedule

INTERVENTIONS:
Behavioral: Centrifugation Distance — To determine optimal distance off-axis, participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 1 minute. Participants received 5 sessions in a 1-week period. Following a 2-week washout period, participants were rotated in a darkened rotary chair booth with 1 ear positioned 7.0 cm off-axis and the other ear positioned on-axis for 1 minute. Participants received 5 sessions in a 1-week period.
Behavioral: Centrifugation Duration — To determine optimal duration, after a two week washout period, participants were rotated off-axis at 3.5 cm (determined to be optimal in Exp 1) for 3 minutes. Participants received 5 sessions in a 1-week period.
Behavioral: Centrifugation Schedule — To determine optimal schedule, after a two week washout period, participants were rotated off-axis at 3.5 cm (determined to be optimal in Exp 1) for 3 minutes (determined to be optimal in Exp 2). Participants received biweekly sessions for a total of 5 sessions.

SUMMARY:
Recent studies suggest that otolith dysfunction is a common finding in individuals with a history of head trauma/blast exposure and/or noise-induced hearing loss. Therefore, otolith dysfunction may be a significant health concern for the Veteran population, and determining optimal intervention strategies for otolith dysfunction is important for VA healthcare. The purpose of this project is to identify optimum stimulus parameters of a novel treatment, off-axis rotation (centrifugation) for otolith dysfunction, in healthy participants.

DETAILED DESCRIPTION:
The primary function of the vestibular (inner ear balance) system is to maintain gaze and postural stability. The vestibular system is comprised of two types of sensory organs (semicircular canals and otolith organs) each with unique contributions to balance.

Vestibular Rehabilitation (VR) is the treatment of choice for patients experiencing dizziness, imbalance, and mobility impairments related to vestibular dysfunction. VR typically includes gaze stability exercises, gait and balance training, and general conditioning. Gaze stability exercises were developed based on the concepts of adaptation and substitution with the goal of improving gaze stability by facilitating vestibular compensation of the semicircular canal-mediated vestibulo-ocular reflex (VOR).

Many factors that might influence recovery, such as the involvement of different vestibular sensory organs (semicircular canals versus otolith organs) have not been examined to determine their impact on recovery. Most studies examining the effectiveness of VR have used only tests of VOR function (caloric and rotational tests) that measure horizontal semicircular canal to determine vestibular loss. Thus, little is known about interventions to facilitate vestibular compensation of the otolith organs.

Recent studies have demonstrated adaptation following otolith organ stimulation using centrifugation (or linear acceleration), but there is no data regarding optimum stimulus parameters. The concept of using centrifugation for otolith adaptation may be similar to using gaze stability exercises for VOR adaptation. Healthy control subjects (n = 5 per experiment) will participate in three separate experiments to determine: (1) the optimum off-axis distance of the rotary chair, (2) the optimum duration of off-axis rotation (OAR), and (3) the optimum OAR stimulation/training schedule.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Documented balance or mobility problems, or healthy control without imbalance
* Otolith dysfunction or healthy control without vestibular dysfunction

Exclusion Criteria:

* Progressive neurological disorders and central vestibular abnormalities
* Benign paroxysmal positional vertigo
* Superior semicircular canal dehiscence
* Middle-ear pathology with conductive hearing loss
* Lower extremity joint replacement
* Cognitive impairment (Mini Mental Status Exam < 24/30)
* Severe depression (geriatric depression scale 10)
* Severe anxiety (geriatric anxiety inventory 11/30)
* Best-corrected visual acuity worse than 20/40 in the better eye

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Hall, PhD PT, Principal Investigator — Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN
Locations (1):
- Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Centrifugation: Each subject will complete training at 3.5 cm off-axis. Participants will be rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis. Subjects will have a wash out period of at least 2 weeks in between chair training distance (3.5 cm or 7.0 cm) until static SVV returns to normal. Then subjects will complete training at 7.0 cm off-axis. Participants will be rotated in a darkened rotary chair booth with 1 ear positioned 7.0 cm off-axis and the other ear positioned on-axis.
  Participants will receive 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo will be assessed at the start and end of each session.
Period: Centrifugation - Distance
Arm/Group | Centrifugation
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Centrifugation - Duration
Arm/Group | Centrifugation
Started | 5
Completed | 5
Not Completed | 0
Period: Centrifugation - Schedule
Arm/Group | Centrifugation
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Centrifugation Distance: Each subject will complete training at both chair positions (3.5 cm off-axis and 7.0 cm off-axis). Subjects will be randomized to start with either chair position (3.5 cm or 7.0 cm) and have a wash out period of at least 2 weeks in between chair training distance (3.5 cm or 7.0 cm) until static SVV returns to normal.
  Participants will be rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm or 7.0 cm off-axis and the other ear positioned on-axis. Participants will receive 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo will be assessed at the start and end of each session.
Arm/Group | Centrifugation Distance
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (3.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
static subjective visual vertical [Mean (Standard Deviation); unit: degrees] — Assesses spatial perception of verticality and is influenced by otolith function. Perception of vertical is measured in a darkened room with subject seated upright.
  degrees | 1.32 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in Static Subjective Visual Vertical (SVV)
Description: Static subjective visual vertical (SVV) assesses spatial perception and is influenced by otolith function. Perception of vertical is measured in a darkened room with subject seated upright. The test assesses an individual's ability to adjust a laser line to be parallel with true vertical in the absence of any other visual cues. The start position of line for SVV testing is randomized and participants are instructed to use the track ball to position the line in a vertical position. Five trials are completed, and the software calculates the distance (in degrees) from vertical. The average of the trials is calculated and used for data analysis.
Time Frame: baseline, immediately after 5 sessions of OAR training (1 week)
Population: The progression through the study is sequential with participants first being tested at 3.5 cm and then at 7.0 cm (both for 1 minute duration) after a two-week washout period. Six participants initiated study testing at 3.5 cm for 1- minute duration, but one participant did not continue with the study. Thus, that participants data are available for the dataset at Distance = 3.5 cm and Duration = 1 minute.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Centrifugation Distance - 3.5 cm: Each subject completed training at chair position of 3.5 cm off-axis.
  Participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 1 minute. Participants received 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo was assessed at the start and end of each session.
- Centrifugation Distance - 7.0 cm: Each subject completed training at chair position of 7.0 cm off-axis after completing training with chair position at 3.5 cm off-axis and having a wash out period of at least 2 weeks (or until static SVV returned to normal) prior to chair training at distance of 7.0 cm.
  Participants were rotated in a darkened rotary chair booth with 1 ear positioned 7.0 cm off-axis and the other ear positioned on-axis for 1 minute. Participants received 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo was assessed at the start and end of each session.
- Centrifugation Duration - 1 Minute: Each subject completed training at chair position of 3.5 cm off-axis.
  Participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 1 minute duration. Participants received 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo was assessed at the start and end of each session.
- Centrifugation Duration - 3 Minutes: After a wash out period of at least 2 weeks (or until static SVV returns to normal), each subject completed training at chair position of 3.5 cm off-axis.
  Participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 3 minutes duration. Participants received 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo was assessed at the start and end of each session.
- Centrifugation Schedule - Daily: After a wash out period of at least 2 weeks (or until static SVV returned to normal), each subject completed training at chair position of 3.5 cm off-axis.
  Participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 3 minutes. Participants received 5 consecutive sessions in a 1-week period (Monday-Friday). Static subjective visual vertigo was assessed at the start and end of each session.
- Centrifugation Schedule - Biweekly: After a wash out period of at least 2 weeks (or until static SVV returned to normal), each subject completed training at chair position of 3.5 cm off-axis.
  Participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 3 minutes. Participants received biweekly sessions for a total of 5 sessions. Static subjective visual vertigo was assessed at the start and end of each session.
Arm/Group | Centrifugation Distance - 3.5 cm | Centrifugation Distance - 7.0 cm | Centrifugation Duration - 1 Minute | Centrifugation Duration - 3 Minutes | Centrifugation Schedule - Daily | Centrifugation Schedule - Biweekly
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 5 | 5
degrees | 0.69 (0.51) | 0.58 (1.47) | 0.69 (0.51) | 0.89 (1.14) | 0.89 (1.14) | 0.32 (1.22)
Statistical Analysis 1: Comparison: Centrifugation Distance - 3.5 cm vs Centrifugation Distance - 7.0 cm; Null hypothesis: The change in SVV (Post-OAR - Pre-OAR) will not be different for the off-axis distance of 3.5 cm and 7.0 cm; Test type: Superiority; p = 0.97, t-test, 2 sided; Paired samples t-test for change in SVV (measured in degrees)
Statistical Analysis 2: Comparison: Centrifugation Duration - 1 Minute vs Centrifugation Duration - 3 Minutes; Null hypothesis: The change in SVV (Post-OAR - Pre-OAR) will not be different for the centrifugation duration of 1 minute and 3 minutes; Test type: Superiority; p = 0.51, t-test, 2 sided; Paired samples t-test for change in SVV (measured in degrees)
Statistical Analysis 3: Comparison: Centrifugation Schedule - Daily vs Centrifugation Schedule - Biweekly; Null hypothesis: The change in SVV (Post-OAR - Pre-OAR) will not be different for the centrifugation schedule of daily OAR and biweekly OAR for a total of 5 sessions; Test type: Superiority; p = 0.44, t-test, 2 sided; Paired samples t-test for change in SVV (measured in degrees)

ADVERSE EVENTS:
Time Frame: Assessment of symptoms was performed immediately following completion of each session of off-axis rotation for a total of 5 sessions within a centrifugation parameter, approximately 3 months.
Description: To assess adverse events following off-axis rotation, participants completed visual analog scales to quantify severity of symptoms (nausea, disorientation, anxiety, imbalance, dizziness).
Groups:
- Centrifugation Distance - 3.5: Participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 1 minute. Participants received 1 daily session for 5 consecutive days.
- Centrifugation Distance - 7.0: Following a washout period of 2 weeks (or until SVV returned to baseline), participants were rotated in a darkened rotary chair booth with 1 ear positioned 7.0 cm off-axis and the other ear positioned on-axis for 1 minute. Participants received 1 daily session for 5 consecutive days.
- Centrifugation Duration - 3 Minutes: Following a washout period of 2 weeks (or until SVV returned to baseline), participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 3 minutes. Participants received 1 daily session for 5 consecutive days.
- Centrifugation Schedule - Biweekly: Following a washout period of 2 weeks (or until SVV returned to baseline), participants were rotated in a darkened rotary chair booth with 1 ear positioned 3.5 cm off-axis and the other ear positioned on-axis for 3 minutes. Participants received biweekly sessions for a total of 5 sessions.
Arm/Group | Centrifugation Distance - 3.5 | Centrifugation Distance - 7.0 | Centrifugation Duration - 3 Minutes | Centrifugation Schedule - Biweekly
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 4/5 | 5/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Centrifugation Distance - 3.5 (N=6) | Centrifugation Distance - 7.0 (N=5) | Centrifugation Duration - 3 Minutes (N=5) | Centrifugation Schedule - Biweekly (N=5)
Symptom of Nausea (General disorders) | 1 (4) | 3 (4) | 3 (8) | 2 (4) — Any increase in symptom (nausea) severity > 0.2 measured using a visual analog scale (Range: 0-10) was included as an adverse event.
Symptom of Disorientation (General disorders) | 6 (17) | 4 (16) | 4 (15) | 4 (10) — Any increase in symptom (disorientation) severity > 0.2 measured using a visual analog scale (Range: 0-10) was included as an adverse event.
Symptom of Anxiety (General disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) — Any increase in symptom (anxiety) severity > 0.2 measured using a visual analog scale (Range: 0-10) was included as an adverse event.
Symptom of Dizziness (General disorders) | 4 (8) | 2 (5) | 3 (7) | 1 (1) — Any increase in symptom (dizziness) severity > 0.2 measured using a visual analog scale (Range: 0-10) was included as an adverse event.
Symptom of Unsteadiness (General disorders) | 4 (9) | 3 (10) | 2 (10) | 1 (5) — Any increase in symptom (unsteadiness) severity > 0.2 measured using a visual analog scale (Range: 0-10) was included as an adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT02652442/Prot_SAP_000.pdf